CLINICAL TRIAL: NCT02701569
Title: Effect of Rebound Therapy on Metabolic Outcomes and Quality of Life in Nigerian Patients With Type 2 Diabetes
Brief Title: Effect of Rebound Exercise in Individuals With Type 2 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of KwaZulu (Other)
Collaborators: Aminu Kano Teaching Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BF389/13
Record Dates: First submitted 2016-02-17; First posted 2016-03-08 (Estimated); Last update posted 2016-10-27 (Estimated); Status verified 2016-02

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Rebound exercise (Experimental): Repeated jumping on a mini trampoline was performed with feet slightly apart
  Interventions: Other: Rebound exercise
- Control (No Intervention): No exercise was administered but participants continued with routine medical care

INTERVENTIONS:
Other: Rebound exercise — Repeated jumping on a mini trampoline was administered
  Other Names: Mini trampoline rebounding
  Arms: Rebound exercise

SUMMARY:
The purpose of this study was to investigate the effect of rebound exercise (mini trampoline jumping) on metabolic outcomes and quality of life in patients with Type 2 Diabetes.

DETAILED DESCRIPTION:
The exercise involved jumping on the mini trampoline with feet slightly apart. Participants stood on the mid portion of the trampoline bed and made repeated up-and-down bouncy movements. Each foot strike equals one step or bounce. With each landing, the mat of the trampoline underwent deformation and the springs released the energy stored in them such that the participant was made to bounce off the mat. Exercise was administered for between 10 - 15 minutes after which a 5-minute period of rest was allowed. A heart rate monitor was used to guide the intensity of the exercise in the moderate range. Each participant accumulated between 20 and 30 minutes of rebound exercise (bouncing on a mini trampoline) per session, administered three times per week for 12 weeks. All data were captured at baseline and at the end of the 12-week intervention period.

ELIGIBILITY:
Inclusion Criteria:

* 30- to 60-year-old male and female individuals;
* A diagnosis of type 2 diabetes ≤ 5 years;
* Attendance at the Diabetes Outpatient Clinics of Aminu Kano Teaching Hospital and Murtala Muhammad Specialist Hospital in Kano, Northwestern Nigeria;
* Self-ambulatory;
* An inactive lifestyle over the last year.

Exclusion Criteria:

* A diagnosis of type 2 diabetes for more than 5 years;
* Hypertension (systolic and diastolic blood pressure more than 140 and 90 mmHg, respectively) or treatment for hypertension;
* Use of insulin therapy
* Lower limb weakness and/or deformities with loss of protective sensation in the feet;
* Back, shoulder or knee problems and/or joint instability;
* History of coronary artery disease, retinopathy and nephropathy;
* Myocardial infarction, cardiac or abdominal surgery within the previous 6 months;
* History of fractures of the spine, hip, knee and/or ankle joints.

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2014-07; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Glycated hemoglobin | 3 months
  Glycated hemoglobin was assessed using the mini-column ion-exchange chromatographic method and expressed in percentage

SECONDARY OUTCOMES:
Fasting plasma glucose | 3 months
  Fasting plasma glucose (in molar concentration) was measured by glucose oxidase assay using a glucose analyzer
Fasting insulin | 3 months
  Fasting insulin (in gravimetric unit) was determined using a commercially available ELISA human insulin kit
High-density lipoprotein cholesterol | 3 months
  High-density lipoprotein cholesterol (in molar concentration) was enzymatically determined using commercial kits
Total cholesterol | 3 months
  Total cholesterol (in molar concentration) was enzymatically determined using commercial kits
Triglycerides | 3 months
  Triglycerides (in molar concentration) were enzymatically determined using commercial kits
Low-density lipoprotein cholesterol | 3 months
  Low-density lipoprotein cholesterol (in molar concentration) was estimated using the Friedewald formula.
Quality of life | 3 months
  The short-form 36 health questionnaire was used to assess participants' quality of life and expressed in percentage
Body mass | 3 months
  Body mass in kilograms was determined using a calibrated weighing scale
Height | 3 months
  Height in meters was determined using a stadiometer
Heart rate | 3 months
  Heart rate was measured in beats per minute using a calibrated electronic device
Respiratory rate | 3 months
  Respiratory rate (in cycles per minute) was measured by observing and counting the number of times the chest rose in one minute
Blood pressure | 3 months
  Blood pressure in millimeters of mercury (mmHg) was measured using a calibrated electronic device
Maximal oxygen consumption | 3 months
  Maximal oxygen consumption in milliliters per kilogram per minute (ml/kg/min) was obtained from exercise stress testing
Diabetes-related emotional distress as measured by the Problem Areas in Diabetes Scale | 3 months
  Diabetes-related emotional distress was expressed in percentage
Well-Being as measured by the World Health Organization-Well-Being Index | 3 months
  Participants' well-being was expressed in percentage
Treatment satisfaction as measured by the World Health Organization-Diabetes Treatment Satisfaction Questionnaire | 3 months
  Score ranges from 0 (very dissatisfied) to 36 (very satisfied)

OTHER OUTCOMES:
Depressive symptoms as measured by the Beck's Depression Inventory | 3 months
  Score ranges from 0 to 63 with 0 to 13 being minimal and 29 to 63 being severe

CONTACTS AND LOCATIONS:
Overall Officials: Sonill S Maharaj, PhD, Study Chair — UKZN

IPD SHARING:
Plan to Share IPD: No
Data would not be shared